CLINICAL TRIAL: NCT03971188
Title: Ligament Reconstruction Tendon Interposition Versus Internal Brace for the Surgical Treatment of Thumb Carpometacarpal Arthritis: a Prospective Randomized Trial Pilot Study
Brief Title: LRTI vs Internal Brace for CMC OA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 010216
Record Dates: First submitted 2019-05-20; First posted 2019-06-03 (Actual); Results first posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Thumb Carpometacarpal Osteoarthritis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internal Brace (Experimental): Patients will undergo Internal Brace procedure for thumb CMC OA.
  Interventions: Procedure: Trapeziectomy with Internal Brace
- LRTI (Active Comparator): Patients will undergo ligament reconstruction tendon interposition (most commonly performed surgery for thumb CMC OA) and serve as control group.
  Interventions: Procedure: Trapeziectomy with Internal Brace

INTERVENTIONS:
Procedure: Trapeziectomy with Internal Brace — Trapeziectomy is performed in standard fashion. Longitudinal traction applied to thumb. Suture anchor with suture tape is inserted into drill hole at radial thumb metacarpal base. A second suture anchor is inserted into a drill hole at the radial base of the index metacarpal such that the suture tape suspends the thumb at the natural groove. Thumb position and tension assessed.

SUMMARY:
Carpometacarpal osteoarthritis (CMC OA) is a prevalent and disabling disease. Trapeziectomy with ligament reconstruction and tendon interposition (LRTI), the most frequently performed procedure for CMC OA, requires prolonged postoperative immobilization which limits patients' abilities to perform Activities of Daily Life (ADLs) and to work. Trapezium excision and internal brace (IB) stabilization is a largely unstudied novel alternative to LRTI which has demonstrated encouraging short-term clinical outcomes and allows an expedited return to work/activity. In this feasibility and pilot grant application, our overall objective is to investigate critical questions to inform the planning of a definitive randomized controlled trial (RCT) comparing IB and LRTI for patients with CMC OA. Our central hypothesis is that a prospective RCT comparing LRTI and IB is feasible, and that IB will produce superior patient-reported outcomes to LRTI at 6 weeks and 3 months with an expedited return to work/activity. Our specific aims are to (1) Establish feasibility of a definitive trial by determining the proportion of eligible subjects who agree to randomized treatment and determining the follow-up retention rate, (2) Estimate effect sizes and variability in outcomes for planning a definitive RCT, and (3) Characterize objective clinical outcomes (thumb range of motion, grip/pinch strength, radiographic outcomes, complications/need for additional surgery, and cost) and to identify differences in return to work/activity following IB and LRTI. To achieve the study's aims, the investigators will randomize 50 patients as they present to the clinics of the 7 Washington University Orthopaedic Hand surgeons to LRTI (control) or IB (experimental). Patients will follow-up at 2 weeks, 4 weeks, 3 months, and 1 year post-operatively. Primary outcomes will be feasibility (randomization rate, follow-up retention rate), and PROMIS scores at 6 weeks and 3 months. Secondary outcomes will be objective clinical outcomes and return to work/activity. Upon completion of the study's aims, the investigators expect to demonstrate that a prospective, randomized trial comparing ligament reconstruction and tendon interposition (LRTI) and internal brace (IB) is feasible, and that patients who undergo IB will have superior short-term patient-reported outcomes to those who undergo LRTI. Furthermore, the study will generate effect size and variability estimates for a definitive, subsequent randomized controlled trial (RCT). Should the objectives for this study be successful, the IB procedure may be readily incorporated into the Hand surgeon's armamentarium as a viable option for the treatment of CMC OA, and the study will provide essential data to support informed, shared decision-making among patients and their physicians.

ELIGIBILITY:
Inclusion Criteria:

* Age >50
* Isolated treatment of CMC arthritis
* No carpal tunnel syndrome (to avoid outcome data confusion)

Exclusion Criteria:

* Patients with thumb metacarpophalangeal hyperextension being addressed surgically
* Patients with concurrent rheumatoid arthritis/inflammatory arthritis
* Patients with history of chronic opioid use

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Washington University & Barnes-Jewish Orthopedic Center in Chesterfield, St Louis, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Barnes-Jewish Center for Advanced Medicine - South County, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were prospectively randomized to LRTI or STS over a 2- year period (December 2019 to December 2021). The enrollment period was prolonged because of the coronavirus disease 2019 pandemic. Potential study participants were identified as they presented to the clinics of five hand surgeons at a single academic medical center.
Pre-assignment Details: Forty-one patients (42 thumbs) agreed to randomization out of a total of 51 patients (52 thumbs) offered participation. One patient had staged bilateral thumb CMC OA surgery one year apart. Ten patients who initially consented to participate subsequently declined; seven decided against randomization and three elected to forego surgery and continue nonsurgical management. A total of 31 patients (32 thumbs) were randomized out of 51 patients (52 thumbs) offered participation.
Units Other Than Participants: thumbs
Period: Overall Study
Arm/Group | Internal Brace | LRTI
Started | 16; 17 thumbs | 15; 15 thumbs
Completed | 16; 17 thumbs | 15; 15 thumbs
Not Completed | 0; 0 thumbs | 0; 0 thumbs

BASELINE CHARACTERISTICS:
Units Other Than Participants: thumbs
Groups:
- Total: Total of all reporting groups
Arm/Group | Internal Brace | LRTI | Total
Number analyzed (Participants) | 16 | 15 | 31
Number analyzed (thumbs) | 17 | 15 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (8) | 61 (8) | 62 (8)
Sex: Female, Male [Count of Units; unit: thumbs]
  Female | 12 | 12 | 24
  Male | 5 | 3 | 8
Race/Ethnicity, Customized [Count of Units; unit: thumbs]
  Race: Black | 0 | 2 | 2
  Race: White | 16 | 13 | 29
  Race: Other | 1 | 0 | 1
Region of Enrollment [Number; unit: thumbs]
  United States | 17 | 15 | 32
Current smoker [Count of Units; unit: thumbs]
  Yes | 1 | 2 | 3
  No | 16 | 13 | 29
Diabetes [Count of Units; unit: thumbs]
  Yes | 3 | 2 | 5
  No | 14 | 13 | 27
Prior ipsilateral hand surgery [Count of Units; unit: thumbs]
  Yes | 4 | 8 | 12
  No | 13 | 7 | 20
Prior contralateral hand surgery [Count of Units; unit: thumbs]
  Yes | 4 | 5 | 9
  No | 13 | 10 | 23
Preoperative Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety Score [Mean (Standard Deviation); unit: T-score] — The PROMIS Anxiety item banks assess self-reported fear, anxious misery, hyperarousal, and somatic symptoms related to arousal. The PROMIS Anxiety Computer Adaptive Test (CAT) was used, in which participant responses guide the system's choice of subsequent items from the full item bank (29 items in total for adults). T-scores were recorded for each participant. A score of 50 is average for the United States general population with a standard deviation of 10. A higher PROMIS T-score represents more anxiety and a worse outcome, with 100 being the highest score.
  T-score | 48 (9) | 51 (10) | 49 (9)
Pre-op PROMIS Depression Score [Mean (Standard Deviation); unit: T-score] — The PROMIS Depression item banks assess self-reported negative mood, views of self, and social cognition, as well as decreased positive affect and engagement. The PROMIS Depression Computer Adaptive Test (CAT) was used, in which participant responses guide the system's choice of subsequent items from the full item bank (28 items in total for adults). T-scores were recorded for each participant. A score of 50 is average for the United States general population with a standard deviation of 10. A higher PROMIS depression T-score represents a worse outcome, with 100 being the highest score.
  T-score | 47 (8) | 46 (10) | 46 (9)
Work status [Count of Participants; unit: Participants]
  Working | 11 | 6 | 17
  Retired | 5 | 9 | 14

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Follow-Up Retention Rate
Description: The investigators will establish feasibility of a definitive trial by determining the proportion of eligible subjects who agree to randomized treatment and determining follow-up retention rate.
Time Frame: 12 months
Measure: Count of Units; unit: thumbs
Units Other Than Participants: thumbs
Arm/Group | Internal Brace | LRTI
Number analyzed (Participants) | 16 | 15
Number analyzed (thumbs) | 17 | 15
thumbs
  3-month follow-up: Yes | 17 | 13
  3-month follow-up: No | 0 | 2
  1-year follow-up: Yes | 17 | 14
  1-year follow-up: No | 0 | 1

2. Primary Outcome: VAS Pain Scores
Description: Visual Analog Scale (VAS) Pain scores will be collected by a member of our team at all visits. These scores will be compared pre-op and at 2 weeks, 4 weeks, 3 months, and 1 year post-op. Scale ranges from 0 to 10 points. For Pain, 0 indicates no pain and 10 indicates maximum pain.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: thumbs
Arm/Group | Internal Brace | LRTI
Number analyzed (Participants) | 16 | 15
Number analyzed (thumbs) | 17 | 15
score on a scale
  Pre-op | 7.4 (1.3) | 7.7 (1.7)
  2 week | 3.9 (2.3) | 2.9 (2.1)
  4 week | 3.1 (2.3) | 1.8 (1.2)
  3 month | 2.5 (2.3) | 1.6 (1.1)
  1 year | 2.4 (2.5) | 2.4 (2.9)

3. Primary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS) Upper Extremity Scores
Description: PROMIS Upper Extremity scores will be collected at all clinic visits on iPad as per standard protocol for all patients presenting to a Washington University Orthopaedic Surgery clinic. These scores will be compared pre-op and at 2 weeks, 4 weeks, 3 months, and 1 year post-op. All PROMIS domain scores are normalized to a mean score of 50 and standard deviation of 10 intending to minimize floor and ceiling effects and ensure the results are readily understood and communicated. A higher score indicates better upper extremity function.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: T-score
Units Other Than Participants: thumbs
Arm/Group | Internal Brace | LRTI
Number analyzed (Participants) | 16 | 15
Number analyzed (thumbs) | 17 | 15
T-score
  Pre-op | 32.7 (4.8) | 36.0 (8.0)
  2 week | 27.0 (4.6) | 29.6 (6.9)
  4 week | 31.7 (5.6) | 35.6 (7.1)
  3 month | 38.6 (7.3) | 42.7 (7.8)
  1 year | 41.5 (9.8) | 46.7 (6.6)

4. Secondary Outcome: Thumb Range of Motion: Thumb IP Joint Extension
Description: Thumb ROM at carpometacarpal, metacarpophalangeal, and interphalangeal joints will be collected by a member of our team at baseline, 4 weeks, 3 months, and 1 year after surgery. These values will be reported in degrees and compared between the two groups.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Degrees
Units Other Than Participants: thumbs
Arm/Group | Internal Brace | LRTI
Number analyzed (Participants) | 16 | 15
Number analyzed (thumbs) | 17 | 15
Degrees
  Pre-op | 18 (12) | 19 (9)
  4 week | 13 (12) | 11 (10)
  3 month | 11 (11) | 21 (10)
  1 year | 17 (14) | 20 (14)

5. Secondary Outcome: Thumb Range of Motion: Thumb IP Joint Flexion
Description: as for outcome 4
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Degrees
Units Other Than Participants: thumbs
Arm/Group | Internal Brace | LRTI
Number analyzed (Participants) | 16 | 15
Number analyzed (thumbs) | 17 | 15
Degrees
  Pre-op | 49 (14) | 44 (17)
  4 week | 41 (14) | 32 (20)
  3 month | 51 (12) | 50 (12)
  1 year | 52 (10) | 56 (13)

6. Secondary Outcome: Thumb Range of Motion: Thumb MCP Joint Extension
Description: as for outcome 4
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Degrees
Units Other Than Participants: thumbs
Arm/Group | Internal Brace | LRTI
Number analyzed (Participants) | 16 | 15
Number analyzed (thumbs) | 17 | 15
Degrees
  Pre-op | 9 (10) | 14 (10)
  4 week | 7 (8) | 5 (6)
  3 month | 9 (11) | 7 (8)
  1 year | 8 (7) | 10 (12)

7. Secondary Outcome: Thumb Range of Motion: Thumb MCP Joint Flexion
Description: as for outcome 4
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Degrees
Units Other Than Participants: thumbs
Arm/Group | Internal Brace | LRTI
Number analyzed (Participants) | 16 | 15
Number analyzed (thumbs) | 17 | 15
Degrees
  Pre-op | 44 (12) | 48 (10)
  4 week | 29 (11) | 22 (11)
  3 month | 32 (11) | 39 (8)
  1 year | 35 (10) | 47 (9)

8. Secondary Outcome: Thumb Range of Motion: Thumb CMC Joint Palmar Abduction
Description: as for outcome 4
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Degrees
Units Other Than Participants: thumbs
Arm/Group | Internal Brace | LRTI
Number analyzed (Participants) | 16 | 15
Number analyzed (thumbs) | 17 | 15
Degrees
  Pre-op | 47 (6) | 40 (11)
  4 week | 47 (4) | 45 (6)
  3 month | 48 (8) | 49 (6)
  1 year | 47 (6) | 50 (5)

9. Secondary Outcome: Thumb Range of Motion: Thumb CMC Joint Palmar Adduction
Description: as for outcome 4
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Degrees
Units Other Than Participants: thumbs
Arm/Group | Internal Brace | LRTI
Number analyzed (Participants) | 16 | 15
Number analyzed (thumbs) | 17 | 15
Degrees
  Pre-op | 16 (10) | 23 (4)
  4 week | 23 (7) | 27 (5)
  3 month | 16 (9) | 21 (4)
  1 year | 19 (6) | 21 (4)

10. Secondary Outcome: Thumb Range of Motion: Thumb CMC Joint Radial Abduction
Description: as for outcome 4
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Degrees
Units Other Than Participants: thumbs
Arm/Group | Internal Brace | LRTI
Number analyzed (Participants) | 16 | 15
Number analyzed (thumbs) | 17 | 15
Degrees
  Pre-op | 45 (6) | 42 (11)
  4 week | 45 (7) | 39 (6)
  3 month | 49 (11) | 42 (9)
  1 year | 45 (10) | 49 (7)

11. Secondary Outcome: Thumb Range of Motion: Thumb CMC Joint Radial Adduction
Description: as for outcome 4
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Degrees
Units Other Than Participants: thumbs
Arm/Group | Internal Brace | LRTI
Number analyzed (Participants) | 16 | 15
Number analyzed (thumbs) | 17 | 15
Degrees
  Pre-op | 15 (11) | 17 (10)
  4 week | 23 (8) | 21 (9)
  3 month | 15 (9) | 17 (9)
  1 year | 18 (8) | 18 (9)

12. Secondary Outcome: Grip Strength
Description: The investigators will record grip strength PRE-OP and POST-OP (all visits except 2 weeks post-op) in both the operative hands. Grip strength will be measured using dynamometer and recorded in pounds (lbs).
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Pounds (lbs)
Units Other Than Participants: thumbs
Arm/Group | Internal Brace | LRTI
Number analyzed (Participants) | 16 | 15
Number analyzed (thumbs) | 17 | 15
Pounds (lbs)
  Pre-op | 37 (17) | 48 (29)
  4 week | 26 (11) | 22 (21)
  3 month | 41 (16) | 46 (24)
  1 year | 56 (17) | 63 (20)

13. Secondary Outcome: Pinch Strength: Lateral Pinch
Description: The investigators will record pinch strength PRE-OP and POST-OP (all visits except 2 weeks post-op) in the operative hand. Pinch strength will be measured using a pinch gauge and recorded in pounds (lbs). For pinch, the investigators will record "lateral/key pinch" AND "3-point pinch."
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Pounds (lbs)
Units Other Than Participants: thumbs
Arm/Group | Internal Brace | LRTI
Number analyzed (Participants) | 16 | 15
Number analyzed (thumbs) | 17 | 15
Pounds (lbs)
  Pre-op | 9 (4) | 11 (6)
  4 week | 5 (3) | 3 (3)
  3 month | 9 (3) | 10 (5)
  1 year | 13 (4) | 13 (5)

14. Secondary Outcome: Pinch Strength: Three-Point Pinch
Description: as for outcome 13
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Pounds (lbs)
Units Other Than Participants: thumbs
Arm/Group | Internal Brace | LRTI
Number analyzed (Participants) | 16 | 15
Number analyzed (thumbs) | 17 | 15
Pounds (lbs)
  Pre-op | 8 (6) | 9 (4)
  4 week | 4 (2) | 2 (3)
  3 month | 7 (3) | 11 (6)
  1 year | 11 (3) | 12 (4)

15. Secondary Outcome: Thumb Metacarpal Radiographic Subsidence: Trapezial Space Ratio Reduction
Description: Posteroanterior wrist and Roberts view C-arm XRs from pre-op, 3 months post-op, and 1 year post-op were obtained. Thumb metacarpal subsidence was calculated using the trapezial space ratio (TSR) measured on a posteroanterior wrist radiograph.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Percent reduction of TSR
Units Other Than Participants: thumbs
Arm/Group | Internal Brace | LRTI
Number analyzed (Participants) | 16 | 15
Number analyzed (thumbs) | 17 | 15
Percent reduction of TSR
  3 months | 48 (22.4) | 42 (13.6)
  1 year | 55 (18.4) | 46 (12.2)

16. Secondary Outcome: Return to Work/Activity
Description: The investigators will track return to work/activity by asking patients at each follow-up visit (1) IF they have returned to their work and baseline activity, and (2) if so, HOW LONG AFTER THEIR SURGERY did they return (ie, 2 weeks, 4 weeks, 6 weeks, 2 mos, 2.5 mos, 3 mos, 4 mos, 5 mos, >6 mos). Return to work and activity will be compared between the two treatment groups.
Time Frame: 12 months
Measure: Count of Units; unit: thumbs
Units Other Than Participants: thumbs
Arm/Group | Internal Brace | LRTI
Number analyzed (Participants) | 16 | 15
Number analyzed (thumbs) | 17 | 15
thumbs
  2 week: Yes | 4 | 7
  2 week: No | 13 | 8
  4 week: Yes | 8 | 9
  4 week: No | 9 | 6
  3 month: Yes | 13 | 14
  3 month: No | 4 | 1
  1 year: Yes | 17 | 15
  1 year: No | 0 | 0

ADVERSE EVENTS:
Time Frame: One year
Description: Mild complications were defined as having minor clinical impact (eg, scar tenderness or sensory disturbances). Moderate complications were defined as clinically relevant with delay in patient recovery but resolved by 1-year and not severe enough to need revision surgery (eg, superficial infections, mild CRPS type I). Severe complications were those that resulted in revision surgery or impaired hand function at 1-year (eg, deep infections requiring irrigation & debridement, severe CRPS type I).
Arm/Group | Internal Brace | LRTI
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/15
Serious Adverse Events (participants affected / at risk) | 1/17 | 0/15
Other Adverse Events (participants affected / at risk) | 4/17 | 1/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Internal Brace (N=17) | LRTI (N=15)
Concern for deep surgical site infection (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — A participant had osteolysis on x-rays with concern for infection, requiring irrigation & debridement and implant removal 9 months from index surgery. Intraoperative cultures were negative for infection, pathology demonstrated chronic inflammation.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Internal Brace (N=17) | LRTI (N=15)
Persistent thumb base pain pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — One of 15 LRTI participants had a mild complication of persistent pain at the thumb base.
Painless first metacarpal osteolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — One participant had painless first metacarpal base osteolysis.
Hypersensitivity of thumb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — One participant had hypersensitivity of the thumb that resolved with gabapentin.
Superficial skin infection (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — One participant had a superficial skin infection that required oral antibiotics.
Fall with wrist injury (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — One participant sustained a fall 2 weeks after surgery resulting in a partial flexor carpi radials tendon injury in the surgical extremity.

LIMITATIONS AND CAVEATS:
First, patients randomized to LRTI and STS participated in different postoperative rehab protocols, which may be a confounding factor in interpreting outcomes. Second, it was not possible to blind surgeons or patients to the procedures and rehab protocol, introducing potential bias. Third, the size of this initial RCT was not sufficient to balance confounding variables between groups. Finally, our cohort was underpowered to detect statistically significant differences in outcome measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-09-09): https://cdn.clinicaltrials.gov/large-docs/88/NCT03971188/Prot_SAP_000.pdf
  • Informed Consent Form (2023-06-19): https://cdn.clinicaltrials.gov/large-docs/88/NCT03971188/ICF_001.pdf